CLINICAL TRIAL: NCT00887198
Title: A Phase 3, Randomized, Double-blind, Placebo-Controlled Study of Abiraterone Acetate (CB7630) Plus Prednisone in Asymptomatic or Mildly Symptomatic Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Abiraterone Acetate in Asymptomatic or Mildly Symptomatic Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016927; COU-AA-302 (Other: Janssen Research & Development, LLC); 2008-008004-41 (EudraCT Number)
Record Dates: First submitted 2009-04-18; First posted 2009-04-23 (Estimated); Results first posted 2015-04-09 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Abiraterone acetate; CB7630; CRPC; Metastatic castration-resistant prostate cancer; hormone refractory prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + prednisone (Placebo Comparator): Placebo plus prednisone
  Interventions: Drug: Placebo; Drug: Prednisone
- Abiraterone + prednisone (Experimental): Abiraterone acetate plus prednisone
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone acetate — 1000 mg per day (4 x 250-mg tablets) taken orally.
  Arms: Abiraterone + prednisone
Drug: Placebo — 4 placebo tablets per day taken orally.
  Arms: Placebo + prednisone
Drug: Prednisone — 5 mg tablet orally twice daily.

SUMMARY:
This is a phase 3 study to compare the clinical benefit of abiraterone acetate plus prednisone with placebo plus prednisone in asymptomatic or mildly symptomatic patients with metastatic castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
This is a randomized (individuals will be assigned by chance to study treatments), double-blind (individuals and study personnel will not know the identity of study treatments), placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial)-controlled study in approximately 1,000 medically or surgically castrated male patients with metastatic CRPC who have shown tumor progression and are asymptomatic or mildly symptomatic. The study period will consist of screening, treatment, and follow-up phases. Patients will receive study treatment (abiraterone acetate or placebo) plus prednisone until radiographic progression of disease and/or unequivocal clinical progression. Efficacy evaluations will be performed throughout the treatment period and safety will be assessed until 30 days after the last dose of abiraterone acetate. throughout the study. Follow-up will continue for up to 60 months (5 years) or until the patient dies, is lost to follow-up, or withdraws informed consent. At the interim analysis of overall survival (OS; 43% of death events), the independent data monitoring committee (IDMC) reviewed the efficacy and safety data and concluded that all of the data pointed to a significant advantage for patients in one arm of the study compared with the other arm thereby unanimously recommending unblinding the study and allowing crossover from the placebo arm to active therapy. Patients currently receiving placebo will be offered crossover therapy to abiraterone acetate. Treatment for patients who were originally randomized to the abiraterone acetate treatment group will not change. Patients will be discontinued from long term follow-up at the time of the Clinical Cut-Off Date for Final Analysis (CCO-FA); however, patients still receiving treatment with abiraterone acetate at the CCO-FA will be offered to receive continued treatment for an additional period of up to 3 years or until disease progression or unacceptable toxicity. For these patients, safety assessment will be performed while continuing treatment, and for 30 days after the last dose of abiraterone acetate.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic castration-resistant prostate cancer (CRPC)
* Previous anti-androgen therapy and progression after withdrawal
* ECOG performance status of either 0 or 1
* Medical or surgical castration with testosterone less than 50 ng/dL
* Life expectancy of at least 6 months

Exclusion Criteria:

* Prior cytotoxic chemotherapy or biologic therapy for CRPC
* Prior ketoconazole for prostate cancer
* Known brain metastasis or visceral organ metastasis
* Use of opiate analgesics for cancer-related pain, including codeine and dextropropoxyphene, currently or anytime within 4 weeks of Cycle 1 Day 1

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1088 (Actual)
Dates: Start 2009-04-28 (Actual); Primary Completion 2014-03-31 (Actual); Study Completion 2017-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (134):
- United States (48):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Bellflower, California
  - Los Angeles, California
  - Marina del Rey, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Stanford, California
  - Aurora, Colorado
  - New Haven, Connecticut
  - Boca Raton, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Kansas City, Kansas
  - Metairie, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Dearborn, Michigan
  - Saint Louis Park, Minnesota
  - St Louis, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - East Syracuse, New York
  - New Hyde Park, New York
  - New York, New York
  - Syracuse, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Canton, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Myrtle Beach, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (19):
  - Adelaide
  - Camperdown
  - Footscray
  - Frankston
  - Garran
  - Geelong
  - Heidelberg
  - Herston
  - Hornsby
  - Kogarah
  - Kurralta Park
  - Lismore
  - Liverpool
  - Malvern
  - Parkville
  - Perth
  - South Brisbane
  - Southport
  - Subiaco
- Belgium (6):
  - Aalst
  - Antwerp
  - Ghent
  - Hasselt
  - Leuven
  - Roeselare
- Canada (10):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- France (9):
  - Caen
  - Clichy
  - Dijon
  - La Roche-sur-Yon
  - Lyon
  - Montpellier
  - Paris
  - Tours
  - Villejuif
- Germany (13):
  - Aachen
  - Berlin
  - Braunschweig
  - Dresden
  - Düsseldorf
  - Hamburg
  - Hanover
  - Homburg
  - Kempen
  - Leipzig
  - München
  - Münster
  - Wuppertal
- Greece (2):
  - Athens
  - Larissa
- Netherlands (4):
  - Amsterdam
  - Heerlen
  - Nijmegen
  - Rotterdam
- Spain (7):
  - A Coruña
  - Barcelona
  - L'Hospitalet de Llobregat
  - Madrid
  - Oviedo
  - Santander
  - Santiago de Compostela
- Sweden (5):
  - Gothenburg
  - Malmo
  - Stockholm
  - Uppsala
  - Vaxjo
- United Kingdom (11):
  - Birmingham
  - Cambridge
  - Glasgow
  - Leeds
  - London
  - Manchester
  - Metropolitan Borough of Wirral
  - Newcastle upon Tyne
  - Oxford
  - Sutton
  - Whitchurch

REFERENCES:
- [Derived] Lorente D, Llacer C, Lozano R, de Velasco G, Romero-Laorden N, Rodrigo M, Sanchez-Iglesias A, di Capua C, Castro E, Ferrer C, Sanchez-Hernandez A, Olmos D. Prognostic Score and Benefit from Abiraterone in First-line Metastatic, Castration-resistant Prostate Cancer. Eur Urol. 2021 Nov;80(5):641-649. doi: 10.1016/j.eururo.2021.07.014. Epub 2021 Aug 6. PMID 34373138
- [Derived] Miller K, Carles J, Gschwend JE, Van Poppel H, Diels J, Brookman-May SD. The Phase 3 COU-AA-302 Study of Abiraterone Acetate Plus Prednisone in Men with Chemotherapy-naive Metastatic Castration-resistant Prostate Cancer: Stratified Analysis Based on Pain, Prostate-specific Antigen, and Gleason Score. Eur Urol. 2018 Jul;74(1):17-23. doi: 10.1016/j.eururo.2017.08.035. Epub 2017 Sep 20. PMID 28939004
- [Derived] de Bono JS, Smith MR, Saad F, Rathkopf DE, Mulders PFA, Small EJ, Shore ND, Fizazi K, De Porre P, Kheoh T, Li J, Todd MB, Ryan CJ, Flaig TW. Subsequent Chemotherapy and Treatment Patterns After Abiraterone Acetate in Patients with Metastatic Castration-resistant Prostate Cancer: Post Hoc Analysis of COU-AA-302. Eur Urol. 2017 Apr;71(4):656-664. doi: 10.1016/j.eururo.2016.06.033. Epub 2016 Jul 9. PMID 27402060
- [Derived] Fizazi K, Flaig TW, Stockle M, Scher HI, de Bono JS, Rathkopf DE, Ryan CJ, Kheoh T, Li J, Todd MB, Griffin TW, Molina A, Ohlmann CH. Does Gleason score at initial diagnosis predict efficacy of abiraterone acetate therapy in patients with metastatic castration-resistant prostate cancer? An analysis of abiraterone acetate phase III trials. Ann Oncol. 2016 Apr;27(4):699-705. doi: 10.1093/annonc/mdv545. Epub 2015 Nov 25. PMID 26609008
- [Derived] Saad F, Shore N, Van Poppel H, Rathkopf DE, Smith MR, de Bono JS, Logothetis CJ, de Souza P, Fizazi K, Mulders PF, Mainwaring P, Hainsworth JD, Beer TM, North S, Fradet Y, Griffin TA, De Porre P, Londhe A, Kheoh T, Small EJ, Scher HI, Molina A, Ryan CJ. Impact of bone-targeted therapies in chemotherapy-naive metastatic castration-resistant prostate cancer patients treated with abiraterone acetate: post hoc analysis of study COU-AA-302. Eur Urol. 2015 Oct;68(4):570-7. doi: 10.1016/j.eururo.2015.04.032. Epub 2015 May 16. PMID 25985882
- [Derived] Xu XS, Ryan CJ, Stuyckens K, Smith MR, Saad F, Griffin TW, Park YC, Yu MK, Vermeulen A, Poggesi I, Nandy P. Correlation between Prostate-Specific Antigen Kinetics and Overall Survival in Abiraterone Acetate-Treated Castration-Resistant Prostate Cancer Patients. Clin Cancer Res. 2015 Jul 15;21(14):3170-7. doi: 10.1158/1078-0432.CCR-14-1549. Epub 2015 Mar 31. PMID 25829400
- [Derived] Morris MJ, Molina A, Small EJ, de Bono JS, Logothetis CJ, Fizazi K, de Souza P, Kantoff PW, Higano CS, Li J, Kheoh T, Larson SM, Matheny SL, Naini V, Burzykowski T, Griffin TW, Scher HI, Ryan CJ. Radiographic progression-free survival as a response biomarker in metastatic castration-resistant prostate cancer: COU-AA-302 results. J Clin Oncol. 2015 Apr 20;33(12):1356-63. doi: 10.1200/JCO.2014.55.3875. Epub 2015 Jan 26. PMID 25624432
- [Derived] Ryan CJ, Smith MR, Fizazi K, Saad F, Mulders PF, Sternberg CN, Miller K, Logothetis CJ, Shore ND, Small EJ, Carles J, Flaig TW, Taplin ME, Higano CS, de Souza P, de Bono JS, Griffin TW, De Porre P, Yu MK, Park YC, Li J, Kheoh T, Naini V, Molina A, Rathkopf DE; COU-AA-302 Investigators. Abiraterone acetate plus prednisone versus placebo plus prednisone in chemotherapy-naive men with metastatic castration-resistant prostate cancer (COU-AA-302): final overall survival analysis of a randomised, double-blind, placebo-controlled phase 3 study. Lancet Oncol. 2015 Feb;16(2):152-60. doi: 10.1016/S1470-2045(14)71205-7. Epub 2015 Jan 16. PMID 25601341
- [Derived] Attard G, de Bono JS, Logothetis CJ, Fizazi K, Mukherjee SD, Joshua AM, Schrijvers D, van den Eertwegh AJ, Li W, Molina A, Griffin TW, Kheoh T, Ricci DS, Zelinsky K, Rathkopf DE, Scher HI, Ryan CJ. Improvements in Radiographic Progression-Free Survival Stratified by ERG Gene Status in Metastatic Castration-Resistant Prostate Cancer Patients Treated with Abiraterone Acetate. Clin Cancer Res. 2015 Apr 1;21(7):1621-7. doi: 10.1158/1078-0432.CCR-14-1961. Epub 2015 Jan 15. PMID 25593303
- [Derived] Aggarwal R, Harris A, Formaker C, Small EJ, Molina A, Griffin TW, Ryan CJ. Response to subsequent docetaxel in a patient cohort with metastatic castration-resistant prostate cancer after abiraterone acetate treatment. Clin Genitourin Cancer. 2014 Oct;12(5):e167-72. doi: 10.1016/j.clgc.2014.03.010. Epub 2014 Mar 28. PMID 24787968
- [Derived] Rathkopf DE, Smith MR, de Bono JS, Logothetis CJ, Shore ND, de Souza P, Fizazi K, Mulders PF, Mainwaring P, Hainsworth JD, Beer TM, North S, Fradet Y, Van Poppel H, Carles J, Flaig TW, Efstathiou E, Yu EY, Higano CS, Taplin ME, Griffin TW, Todd MB, Yu MK, Park YC, Kheoh T, Small EJ, Scher HI, Molina A, Ryan CJ, Saad F. Updated interim efficacy analysis and long-term safety of abiraterone acetate in metastatic castration-resistant prostate cancer patients without prior chemotherapy (COU-AA-302). Eur Urol. 2014 Nov;66(5):815-25. doi: 10.1016/j.eururo.2014.02.056. Epub 2014 Mar 6. PMID 24647231
- [Derived] Basch E, Autio K, Ryan CJ, Mulders P, Shore N, Kheoh T, Fizazi K, Logothetis CJ, Rathkopf D, Smith MR, Mainwaring PN, Hao Y, Griffin T, Li S, Meyers ML, Molina A, Cleeland C. Abiraterone acetate plus prednisone versus prednisone alone in chemotherapy-naive men with metastatic castration-resistant prostate cancer: patient-reported outcome results of a randomised phase 3 trial. Lancet Oncol. 2013 Nov;14(12):1193-9. doi: 10.1016/S1470-2045(13)70424-8. Epub 2013 Sep 25. PMID 24075621
- [Derived] Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, Fizazi K, Mainwaring P, Piulats JM, Ng S, Carles J, Mulders PF, Basch E, Small EJ, Saad F, Schrijvers D, Van Poppel H, Mukherjee SD, Suttmann H, Gerritsen WR, Flaig TW, George DJ, Yu EY, Efstathiou E, Pantuck A, Winquist E, Higano CS, Taplin ME, Park Y, Kheoh T, Griffin T, Scher HI, Rathkopf DE; COU-AA-302 Investigators. Abiraterone in metastatic prostate cancer without previous chemotherapy. N Engl J Med. 2013 Jan 10;368(2):138-48. doi: 10.1056/NEJMoa1209096. Epub 2012 Dec 10. PMID 23228172

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Acetate + Prednisone (AAP): Participants received 1000 milligram (mg) abiraterone acetate tablets (as 4*250 mg tablets) orally once daily along with prednisone 5 mg tablet orally twice daily, from Day 1, Cycle1 (each cycle consist of 28 days) up to radiographic progression of disease and/or unequivocal clinical progression.
- Placebo: Participants received placebo matched to abiraterone acetate tablets orally once daily along with prednisone 5 mg tablet orally twice daily, from Day 1, Cycle1 (each cycle consist of 28 days) up to radiographic progression of disease and/or unequivocal clinical progression.
- Placebo to AA: Participants who were originally assigned to placebo were later on switched to 1,000 milligram (mg) abiraterone acetate tablet (as 4*250 mg tablets) along with prednisone 5 mg tablet.
Period: Randomized Period
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo | Placebo to AA
Started | 546 | 542 | 0
Treated | 542 | 540 | 0
Completed | 0 | 0 | 0
Not Completed | 546 | 542 | 0
Not completed — Ongoing | 42 | 0 | 0
Not completed — Adverse Event | 50 | 33 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Cross-over to AA (under amendment 3) | 0 | 51 | 0
Not completed — Withdrawal by Subject | 41 | 56 | 0
Not completed — Progressive disease | 366 | 370 | 0
Not completed — Other | 42 | 30 | 0
Not completed — Randomized, Not treated | 4 | 2 | 0
Period: Cross Over (Placebo to AA)
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo | Placebo to AA
Started | 0 | 0 | 93 (93= 51 participants(crossed over under amendment 3)+42 participants (crossed over under amendment 4))
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 93
Not completed — Started other prostate cancer treatment | 0 | 0 | 8
Not completed — Ongoing | 0 | 0 | 35
Not completed — Adverse Event | 0 | 0 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Progressive disease | 0 | 0 | 20
Not completed — Other | 0 | 0 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo | Total
Number analyzed (Participants) | 546 | 542 | 1088
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (8.8) | 70.1 (8.72) | 70.3 (8.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 546 | 542 | 1088
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 60 | 72 | 132
  Belgium | 25 | 17 | 42
  Canada | 63 | 37 | 100
  France | 24 | 29 | 53
  Germany | 46 | 32 | 78
  Greece | 7 | 7 | 14
  Italy | 1 | 6 | 7
  Netherlands | 15 | 15 | 30
  Spain | 25 | 20 | 45
  Sweden | 4 | 13 | 17
  United Kingdom | 42 | 56 | 98
  United States | 234 | 238 | 472

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from randomization to date of death from any cause.
Time Frame: From randomization (Day 1) up to end of study (Month 60)
Population: Intent-to-treat (ITT) population included all the randomized participants who were classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo
Number analyzed (Participants) | 546 | 542
Months | 34.66 [32.72 to 36.80] | 30.29 [28.65 to 33.28]

2. Primary Outcome: Radiographic Progression-free Survival (rPFS)
Description: The rPFS was defined as the time from randomization to the occurrence of one of the following: 1) a participant was considered to have progressed by bone scan if - a) the first bone scan with greater than or equal to (>=) 2 new lesions compared to baseline was observed in less than (<) 12 weeks from randomization and was confirmed by a second bone scan taken >=6 weeks later showing >=2 additional new lesions (a total of >=4 new lesions compared to baseline), b) the first bone scan with >=2 new lesions compared to baseline was observed in >=12 weeks from randomization and the new lesions were verified on the next bone scan >=6 weeks later (a total of >=2 new lesions compared to baseline); 2) progression of soft tissue lesions measured by computerized tomography (CT) or magnetic resonance imaging (MRI); 3) death from any cause.
Time Frame: From randomization (Day 1) up to first radiographic progression or cutoff date (Month 18)
Population: ITT population included all the randomized participants who were classified according to their assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo
Number analyzed (Participants) | 546 | 542
Months | NA [11.66 to NA] — Data was not estimable due to insufficient number of participants who had the event. | 8.28 [8.12 to 8.54]

3. Secondary Outcome: Time to Opiate Use for Prostate Cancer Pain
Description: The time interval from the date of randomization to the date of opiate use for cancer pain. Participants who have no opiate use at the time of analysis were censored at the last known date of no opiate use for cancer pain. Participants with no assessment were censored at the date of randomization.
Time Frame: From randomization (Day 1) up to first opiate use or end of study (Month 60)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo
Number analyzed (Participants) | 546 | 542
Months | 33.38 [30.23 to 39.75] | 23.39 [20.27 to 27.53]

4. Secondary Outcome: Time to Initiation of Cytotoxic Chemotherapy
Description: The time interval from the date of randomization to the date of initiation of cytotoxic chemotherapy for prostate cancer. Participants who had no cytotoxic chemotherapy administration at the time of analysis were censored at the last known date when no cytotoxic chemotherapy was administered. Participants with no assessment were censored at the date of randomization.
Time Frame: From randomization (Day 1) up to initiation of cytotoxic chemotherapy or cutoff date (Month 18)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo
Number analyzed (Participants) | 546 | 542
Months | 25.17 [23.26 to NA] — Upper limit was not estimable due to insufficient number of participants who had the event. | 16.82 [14.55 to 19.38]

5. Secondary Outcome: Time to Deterioration in Eastern Cooperative Oncology Group (ECOG) Performance Score by >=1 Point
Description: The time interval from the date of randomization to the first date at which there was at least a 1 grade change (worsening) in the ECOG performance status grade. Participants who had no deterioration in ECOG performance status grade at the time of the analysis were censored at the last known date of no deterioration. ECOG is a 5-point scale, where 0=Fully active, 1=Ambulatory, carry out work of sedentary nature, 2=Ambulatory, capable of all self-care, 3=Capable of limited self-care, confined to bed or chair more than 50% of waking hours, 4=Completely disabled, no self-care, totally confined to bed or chair, 5=Dead. Participants with no assessment were censored at the date of randomization.
Time Frame: From randomization (Day 1) up to first radiographic progression or cutoff date (Month 18)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo
Number analyzed (Participants) | 546 | 542
Months | 12.29 [11.33 to 14.29] | 10.87 [9.49 to 11.76]

6. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: The time interval from the date of randomization to the date of PSA progression as defined in the protocol-specific prostate cancer Working Group 2 (PCWG2) criteria. A participant was considered to have a PSA progression if the PSA level had a 25 percent (%) or greater increase from nadir and an absolute increase of 2 nanogram/milliliter ((ng/mL) or more, which is confirmed by a second value obtained in 3 or more weeks. Participants who had no PSA progression at the time of the analysis were censored at the last known date of no PSA progression. Participants with no on-study PSA assessment or no baseline PSA assessment were censored at the date of randomization.
Time Frame: From randomization (Day 1) up to date of PSA progerssion or cutoff date (Month 18)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo
Number analyzed (Participants) | 546 | 542
Months | 11.07 [8.51 to 11.24] | 5.55 [5.39 to 5.59]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between administration of study drug and up to 30 days after last dose of study drug that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug
Population: Safety analysis set included all participants in the randomized population who received any study drug.
Measure: Number; unit: Participants
Groups:
- Placebo to Abiraterone Acetate: Participants received initially placebo along with prednisone 5 mg tablet, orally, later on switched to 1,000 milligram (mg) abiraterone acetate tablet (as 4*250 mg tablets) along with prednisone 5 mg tablet due to disease progression.
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo | Placebo to Abiraterone Acetate
Number analyzed (Participants) | 542 | 540 | 93
Participants
  With Treatment-Emergent Adverse Events | 541 | 524 | 93
  With Treatment-Emergent Serious Adverse Events | 208 | 148 | 39

8. Secondary Outcome: Mean Plasma Concentrations of Abiraterone
Time Frame: Up to Cycle 5, Day 1
Population: Data was not reported as non-compartmental analysis was not performed due to sparse sampling.
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Maximum Plasma Concentrations of Abiraterone
Time Frame: Up to Cycle 5, Day 1
Population: Data was not reported as non-compartmental analysis was not performed due to sparse sampling.
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Time the Last Quantifiable Concentration of Abiraterone (AUC[0-infinity])
Description: The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Time Frame: Up to Cycle 5, Day 1
Population: Data was not reported as non-compartmental analysis was not performed due to sparse sampling.
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Elimination Half-Life (t1/2)
Description: The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Time Frame: Up to Cycle 5, Day 1
Population: Data was not reported as non-compartmental analysis was not performed due to sparse sampling.
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug (Approximately 5 years)
Description: Safety analysis set included all participants in the randomized population who received any study drug.
Arm/Group | Abiraterone Acetate + Prednisone (AAP) | Placebo | Placebo to AA
Serious Adverse Events (participants affected / at risk) | 215/542 | 156/540 | 40/93
Other Adverse Events (participants affected / at risk) | 530/542 | 505/540 | 86/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate + Prednisone (AAP) (N=542) | Placebo (N=540) | Placebo to AA (N=93)
Anaemia (Blood and lymphatic system disorders) | 8 | 6 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 2
Malaise (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 3 | 3 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 0
Bronchopneumonia (Infections and infestations) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 2 | 3 | 2
Cystitis (Infections and infestations) | 3 | 0 | 0
Gastroenteritis (Infections and infestations) | 6 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 10 | 4 | 1
Pyelonephritis (Infections and infestations) | 3 | 2 | 1
Sepsis (Infections and infestations) | 7 | 2 | 1
Sinusitis (Infections and infestations) | 2 | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 3 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 1
Colonoscopy (Investigations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 0 | 0
Paraparesis (Nervous system disorders) | 1 | 0 | 0
Paraplegia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0
Quadriparesis (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 6 | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 11 | 5 | 3
Hydronephrosis (Renal and urinary disorders) | 2 | 4 | 0
Nephrolithiasis (Renal and urinary disorders) | 3 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 2 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Chemotherapy (Surgical and medical procedures) | 1 | 0 | 0
Pancreatectomy (Surgical and medical procedures) | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 3 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 1
Angina Pectoris (Cardiac disorders) | 6 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 11 | 8 | 0
Atrioventricular Block (Cardiac disorders) | 1 | 1 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 0 | 1
Bifascicular Block (Cardiac disorders) | 1 | 0 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 2 | 0
Cardiac Disorder (Cardiac disorders) | 1 | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 3 | 0 | 0
Conduction Disorder (Cardiac disorders) | 1 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 4 | 1 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 4 | 5 | 2
Myocardial Ischaemia (Cardiac disorders) | 2 | 0 | 0
Supraventricular Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 2 | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 3 | 5 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0
Diverticular Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum Intestinal (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Enterovesical Fistula (Gastrointestinal disorders) | 1 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis Erosive (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal Necrosis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 1 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Oesophageal Mass (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic Disorder (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis Necrotising (Gastrointestinal disorders) | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Varices Oesophageal (Gastrointestinal disorders) | 0 | 1 | 0
Catheter Related Complication (General disorders) | 1 | 0 | 0
Chest Pain (General disorders) | 0 | 1 | 1
Death (General disorders) | 1 | 0 | 0
Disease Progression (General disorders) | 8 | 4 | 6
Gait Disturbance (General disorders) | 1 | 1 | 0
General Physical Health Deterioration (General disorders) | 7 | 2 | 0
Hypothermia (General disorders) | 1 | 0 | 0
Mucosal Inflammation (General disorders) | 1 | 0 | 0
Multi-Organ Failure (General disorders) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 4 | 1
Oedema Peripheral (General disorders) | 2 | 0 | 0
Performance Status Decreased (General disorders) | 0 | 1 | 0
Systemic Inflammatory Response Syndrome (General disorders) | 0 | 0 | 1
Bile Duct Obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Anal Abscess (Infections and infestations) | 0 | 1 | 0
Arthritis Bacterial (Infections and infestations) | 1 | 0 | 0
Biliary Sepsis (Infections and infestations) | 0 | 1 | 0
Bursitis Infective (Infections and infestations) | 1 | 0 | 0
Campylobacter Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Enterococcal Infection (Infections and infestations) | 1 | 0 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Febrile Infection (Infections and infestations) | 0 | 1 | 0
Gallbladder Abscess (Infections and infestations) | 0 | 1 | 0
Gastroenteritis Salmonella (Infections and infestations) | 1 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 1 | 0 | 0
Gingival Infection (Infections and infestations) | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 1 | 0 | 0
Infected Skin Ulcer (Infections and infestations) | 1 | 0 | 0
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 1 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0
Lung Infection (Infections and infestations) | 3 | 0 | 0
Necrotising Fasciitis (Infections and infestations) | 0 | 1 | 0
Parainfluenzae Virus Infection (Infections and infestations) | 1 | 0 | 0
Pneumonia Influenzal (Infections and infestations) | 1 | 1 | 0
Pneumonia Staphylococcal (Infections and infestations) | 1 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 0 | 0
Pseudomonal Bacteraemia (Infections and infestations) | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 3 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 14 | 4 | 5
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 1 | 0
Viral Infection (Infections and infestations) | 1 | 1 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 1
Animal Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Bladder Perforation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cataract Operation Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cystitis Radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Device Dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Gastroenteritis Radiation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 1 | 0 | 0
Implantable Defibrillator Malfunction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Multiple Injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0
Narcotic Intoxication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pubic Rami Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Scapula Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skeletal Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skull Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stress Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 2
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 5 | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 3 | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 0
Blood Uric Acid Increased (Investigations) | 1 | 0 | 0
Electrocardiogram QT Prolonged (Investigations) | 1 | 0 | 0
Electrocardiogram St Segment Depression (Investigations) | 1 | 0 | 0
Lipase Increased (Investigations) | 2 | 0 | 0
Platelet Count Decreased (Investigations) | 1 | 0 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 2 | 0 | 0
Fluid Retention (Metabolism and nutrition disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 4 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Jaw Cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
B-Cell Type Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Central Nervous System Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Intestinal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Malignant Neoplasm of Ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastatic Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Urethral Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 1 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 2 | 0
Cerebral Ischaemia (Nervous system disorders) | 3 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 6 | 2 | 0
Embolic Stroke (Nervous system disorders) | 1 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 1 | 0 | 0
Memory Impairment (Nervous system disorders) | 0 | 1 | 0
Migraine with Aura (Nervous system disorders) | 0 | 1 | 0
Nerve Root Compression (Nervous system disorders) | 2 | 0 | 1
Neurological Symptom (Nervous system disorders) | 1 | 0 | 0
Spinal Cord Compression (Nervous system disorders) | 7 | 4 | 0
Syncope Vasovagal (Nervous system disorders) | 2 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0 | 0
Confusional State (Psychiatric disorders) | 1 | 2 | 0
Bladder Mass (Renal and urinary disorders) | 1 | 0 | 0
Bladder Obstruction (Renal and urinary disorders) | 1 | 1 | 0
Bladder Spasm (Renal and urinary disorders) | 0 | 1 | 0
Bladder Tamponade (Renal and urinary disorders) | 1 | 0 | 0
Calculus Bladder (Renal and urinary disorders) | 0 | 0 | 2
Calculus Ureteric (Renal and urinary disorders) | 2 | 0 | 0
Haemorrhage Urinary Tract (Renal and urinary disorders) | 1 | 0 | 0
Obstructive Uropathy (Renal and urinary disorders) | 0 | 2 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 3 | 0
Renal Failure Acute (Renal and urinary disorders) | 3 | 2 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 0 | 0
Ureteric Obstruction (Renal and urinary disorders) | 2 | 2 | 0
Ureteric Stenosis (Renal and urinary disorders) | 0 | 1 | 0
Urethral Obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urethral Stenosis (Renal and urinary disorders) | 0 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 6 | 3 | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 1 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatic Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Scrotal Pain (Reproductive system and breast disorders) | 0 | 1 | 0
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 12 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Tonsillar Cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Aortic Valve Replacement (Surgical and medical procedures) | 1 | 0 | 0
Knee Arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
Transurethral Prostatectomy (Surgical and medical procedures) | 0 | 1 | 0
Arterial Thrombosis (Vascular disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 4 | 2 | 0
Embolism Venous (Vascular disorders) | 1 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 1 | 0
Peripheral Embolism (Vascular disorders) | 0 | 1 | 0
Peripheral Vascular Disorder (Vascular disorders) | 1 | 0 | 0
Venous Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate + Prednisone (AAP) (N=542) | Placebo (N=540) | Placebo to AA (N=93)
Anaemia (Blood and lymphatic system disorders) | 59 | 53 | 12
Constipation (Gastrointestinal disorders) | 144 | 112 | 15
Diarrhoea (Gastrointestinal disorders) | 135 | 98 | 13
Dyspepsia (Gastrointestinal disorders) | 62 | 28 | 1
Nausea (Gastrointestinal disorders) | 144 | 127 | 15
Vomiting (Gastrointestinal disorders) | 86 | 61 | 12
Asthenia (General disorders) | 46 | 46 | 1
Fatigue (General disorders) | 243 | 200 | 27
Pyrexia (General disorders) | 54 | 33 | 5
Bronchitis (Infections and infestations) | 34 | 14 | 0
Nasopharyngitis (Infections and infestations) | 65 | 46 | 5
Sinusitis (Infections and infestations) | 29 | 5 | 3
Contusion (Injury, poisoning and procedural complications) | 81 | 49 | 6
Fall (Injury, poisoning and procedural complications) | 47 | 20 | 12
Anorexia (Metabolism and nutrition disorders) | 56 | 40 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 52 | 41 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 99 | 68 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 14 | 15 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 172 | 131 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 40 | 32 | 3
Dizziness (Nervous system disorders) | 81 | 73 | 7
Headache (Nervous system disorders) | 86 | 66 | 9
Anxiety (Psychiatric disorders) | 30 | 23 | 4
Depression (Psychiatric disorders) | 32 | 19 | 3
Insomnia (Psychiatric disorders) | 82 | 62 | 5
Haematuria (Renal and urinary disorders) | 56 | 32 | 4
Nocturia (Renal and urinary disorders) | 38 | 29 | 0
Pollakiuria (Renal and urinary disorders) | 56 | 55 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 106 | 74 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 71 | 52 | 7
Rash (Skin and subcutaneous tissue disorders) | 49 | 21 | 1
Hypertension (Vascular disorders) | 129 | 73 | 6
Abdominal Pain (Gastrointestinal disorders) | 49 | 44 | 5
Oedema Peripheral (General disorders) | 148 | 119 | 22
Lower Respiratory Tract Infection (Infections and infestations) | 12 | 13 | 5
Upper Respiratory Tract Infection (Infections and infestations) | 74 | 43 | 4
Urinary Tract Infection (Infections and infestations) | 49 | 40 | 11
Skin Laceration (Injury, poisoning and procedural complications) | 13 | 15 | 6
Alanine Aminotransferase Increased (Investigations) | 70 | 26 | 3
Aspartate Aminotransferase Increased (Investigations) | 63 | 25 | 4
Weight Decreased (Investigations) | 42 | 27 | 6
Weight Increased (Investigations) | 29 | 40 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 28 | 30 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 199 | 180 | 26
Bone Pain (Musculoskeletal and connective tissue disorders) | 144 | 112 | 14
Groin Pain (Musculoskeletal and connective tissue disorders) | 41 | 22 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 78 | 111 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 35 | 42 | 5
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 97 | 77 | 12
Neck Pain (Musculoskeletal and connective tissue disorders) | 30 | 17 | 2
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 107 | 89 | 16
Neuropathy Peripheral (Nervous system disorders) | 12 | 6 | 7
Urinary Incontinence (Renal and urinary disorders) | 37 | 25 | 0
Hot Flush (Vascular disorders) | 124 | 100 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the Sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.